CLINICAL TRIAL: NCT03707405
Title: Compare the Effectiveness of Modified Toy Cars Training With Various Intensity of Postural Combinations on Mobility and Socialization in Toddlers With Motor Disabilities: a Randomized Controlled Trial.
Brief Title: Compare the Effectiveness of Modified Toy Cars Training With Various Intensity of Postural Combinations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Hsiang-Han Huang, Assistant Professor, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 107WFD2610149
Record Dates: First submitted 2018-07-26; First posted 2018-10-16 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2022-03

CONDITIONS: Young Children With Motor Disabilities
MeSH Terms: interventions — Sitting Position

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- ROC-sit (Active Comparator): Ride-On Cars with Sitting Posture (ROC-sit) The 2-hour training session is composed of a 70-minute driving session and a 40-to-50-minute natural play session, with a 10-mintue break if necessary. The natural play session can be divided into two 20-to-25 sessions depending on the participant's condition. Training will concentrate on building the concept of casual-effect on the switch and car motion, practicing goal-oriented driving (e.g., driving 200 meters and reach for a toy or contact with a person) in public spaces (e.g., hallways, convenient stores, garden, museum) and upper limb use in functional tasks with driving, facilitating hand use in functional tasks for exploration and applying motor skills for mobility and socialization in natural play session. All the programs will be discussed by the family, the treating therapist and the research team.
  Interventions: Behavioral: Ride-On Cars Training with Different Postures
- ROC-sit45 and stand25 (Active Comparator): Ride-On Cars with 45-min Sitting and 25-min Standing Postures (ROC-sit45 and stand25) The training guidelines and time are the same as the ROC-sit group, except for the posture of driving. The 70-minute driving session begins with a 45-minute driving with sitting posture and then transfers to the standing posture for driving 25 minutes.
  Interventions: Behavioral: Ride-On Cars Training with Different Postures
- ROC-sit25 and stand45 (Active Comparator): Ride-On Cars with 25-min Sitting and 45-min Standing Postures (ROC-sit25 and stand45) The training guidelines and time are the same as the ROC-sit group, except for the posture of driving. The 70-minute driving session begins with a 25-minute driving with sitting posture and then transfers to the standing posture for driving 45 minutes.
  Interventions: Behavioral: Ride-On Cars Training with Different Postures
- ROC-stand (Active Comparator): Ride-On Cars with Standing Postures (ROC-stand) The training guidelines and time are the same as the ROC-sit group, except for the posture of driving. The 70-minute standing session can be divided into two 30-minute sessions with 10-minute break, depending on the child's condition with the standing posture.
  Interventions: Behavioral: Ride-On Cars Training with Different Postures

INTERVENTIONS:
Behavioral: Ride-On Cars Training with Different Postures — All programs will include 120 minutes/per session, 2 sessions/per week. All participants will continue their regular therapy during the whole study. The treatment strategy of ROC training with different postures will be based on the exploratory learning which focuses on providing opportunities to the participants to explore environmental properties with various motor patterns during the intervention.
  Other Names: Ride-On Cars with 45-min Sitting and 25-min Standing Postures; Ride-On Cars with 25-min Sitting and 45-min Standing Postures; Ride-On Cars with Standing Postures

SUMMARY:
The three purposes of this study are: 1) to determine the feasibility of applying two types of postural combinations for the ride-on car (ROC) use; 2) to compare the effectiveness of ROC training with various intensity of postural combinations on mobility, socialization and energy expenditure in toddlers with disabilities; and 3) to examine the effects of using the different modes of ROC training (different intensity of postural combinations) on the ICF functioning levels, family perceptions and participation. Modified ride-on toy cars (ROCs) as a type of PMDs have become an innovative, alternative option to enhance independent mobility and socialization in young children with disabilities. Evidence suggested that dose-response effect and energy expenditure of the two postures used for training may result in the observed differences. Therefore, this study is further to examine the effectiveness of ROC training with various intensity of postural combinations on independent mobility, socialization, motivation, physical activity and overall development through low-cost, family-centered approach.

Based on the power analysis from the preliminary results, the investigators will recruit 92 children with disabilities who are between 1 to 3 years old and diagnosed as motor delay (>1.5 sd). They will be randomly assigned to one of the following four groups: ROC-sit group (n=23), ROC-stand group (n=23), ROC training with 45-min sitting and 25-min standing (n=23), and the ROC training group with 25-min sitting and 45-min standing (n=23). The whole study duration will be 24 weeks, including 12-week intervention and 12-week follow-up; the total amount of treatment will be equal for the four groups. Standardized assessments are provided for a total three times, including the time before and after the intervention and in the end of the follow-up phase. All programs will include 120 minutes/per session, 2 sessions/per week. The research team will provide 90-min behavioral videotaping once/per week and let participants wear three accelerometers throughout the 2-hour training. Assessments include mobility, socialization, behavioral coding, family perception and participation. The findings of this study will provide a novel application of ROC training with various intensity of postural combinations on advancing children's mobility, socialization, development and family participation.

DETAILED DESCRIPTION:
Some studies showed the use of laboratory-designed PMDs or modified ride-on cars (ROCs) might increase the child's independent mobility and motivation to master interpersonal tasks and result in positive changes on social functioning.

Modified ROCs as a type of PMDs have become an innovative, alternative option to enhance independent mobility in children with disabilities. Studies have found that the novel application of modified ROCs in home-based, community-based or hospital-based environments might enhance independent mobility, motivation, and social function in young children with motor disabilities. In addition, these studies have indicated that the application of modified ROCs integrating the concept of family-centered service may be beneficial for improving young children's motivation due to their persistence on driving and increased pleasure during training.

The dose-response effect of the ROC use with different postures on mobility function may be the reason relating to the previous findings. The progress of mobility function might be affected due to the focus on increasing socialization over mobility. Moreover, several studies have demonstrated that walking or standing may result in more energy expenditure than other postures, e.g., sitting or lying for children with disabilities. The ROC-stand training group required a total dynamic standing time of 60 to 70 minutes for driving and exploration during each session, which may increase the children's energy expenditure and result in less strength and endurance to move without the ROC. However, the standing posture may provide more opportunities and visual information for children to interact with other people and distal events, which relates to the development of socialization. With these outcomes and possible explanations, the investigators propose that the subsequent research may identify the "dose-response" effect of different postural combinations for the ROC use on mobility and social functions in toddlers with motor disabilities.

In this study, the investigators will modify two types of ride-on toy cars for toddlers with disabilities for the use in the public spaces in the university as part of a 24-week power mobility training program. In addition, the investigators will compare the effectiveness of different intensity of postural combinations for the ROC training on mobility and socialization in toddlers with motor disabilities. The previous 2-hour ROC-training program included an average of 60-to-70-miniute driving (unstructured) and 50-minute natural play (structured) which involved exploration and motor skills training related to mobility and social impairments, such as postural stability, postural control, and social engagement. Based on the previous evidence, the investigators propose two groups which involve different intensity of postural combinations for the ROC use, i.e., one group of 45-minute sitting and 25-minute standing and the other group of 25-minute sitting and 45-minute standing, may be optimal for toddlers with motor disabilities to meet the physical activity guidelines. the investigators further propose these postural combinations of the ROC use may have different effects on mobility and social function, compared to the original use with only one posture. A 4-group comparison design of decreased intensity of sitting posture and increased intensity of standing posture for the ROCs use may provide us a complete examination on the topic of dose-response effect on toddlers with disabilities. In addition, the investigators will examine whether the effects of increased independent mobility and socialization will affect toddler's function on the 3 International Classification of Function (ICF) domains. If our results are generally positive and show significant differences on independent mobility and socialization among the ROC training programs with two different postures and various intensity, it will provide us some alternative ways to improve independent mobility and socialization depending on children's and family's needs.

The specific aims of this study are: 1) to determine the feasibility and examine the effects of ROC training with various intensity of postural combinations on mobility and socialization in toddlers with disabilities; 2) to objectively quantify the intensity and energy expenditure of postural combinations for the ROCs use through accelerometers; 3) to determine the effects of using the different modes of ROC training (different intensity of postural combinations) on the ICF functioning levels, family perceptions and participation.

Method Study Design: A multiple group pretest-posttest control group design will be applied. Four groups will be involved in this project: ride-on car with sitting posture (ROC-sit), ride-on car with standing posture (ROC-stand), and two groups of ride-on car with mixed postures, including one group of 45-min sitting and 25-min standing postures (ROC-sit45 and stand25) and the other group of 25-min sitting and 45-min standing postures (ROC-sit25 and stand45). The study duration for each participant is 24 weeks, including 12-week intervention and 12-week follow-up.

Participants: Participants in the study will be 92 toddlers ages 12 months to 36 months with motor delays. They will be randomly assigned to either the ROC-sit group (23 toddlers), the ROC-stand group (23 toddlers), the ROC-sit45 and stand25 group (23 toddlers) or the ROC-sit25 and stand45 group (23 toddlers). The age group of infants/preschool children is selected based on the previous studies of ROC training in young children with motor disabilities.

Recruitment: The participants will be recruited from self-referrals, health care practitioners, or the hospitals in Taipei or Taoyuan where toddlers with motor delays are receiving outpatient rehabilitations. The research team will initially post flyers describing the study at clinical settings and contact the therapists in the clinical settings to introduce the goals, criteria and general procedure of the study. Parents/guardians will obtain information about the study through the flyers and their therapists. The research team will contact the parent/guardian to explain study details and provide them the opportunity to ask questions. Children of parents/guardians who provide informed consent will participate in the study.

Procedure: Each participant of the ride-on car training groups will have either a customized, sitting-style toy car or a standing-style toy car, depending on the assigned group. The adaptations are all assembled by PVC pipes which can be adjusted easily during each training session. After modifications, they will receive pre-intervention measurements, including developmental assessments, behavioral videotaping and self-developed questionnaires. The self-developed questionnaires were designed to examine parental perceptions on the PMDs use and children's capabilities in the previous studies. The pretest and posttest developmental assessments and questionnaires will be completed in a testing room at Chang Gung University by a licensed occupational therapist who is blinded to the study purpose and not involved in the treatment. These assessments will occur on three occasions: before and after the 12-week intervention (T1 & T2) and the end of the 12-week follow-up phase (T3). During the 12-week intervention, the locomotion (i.e., driving) and socialization behaviors for the four ROC training groups will also be videotaped by the research team for 1.5 hours during one session/per week at the university. In addition, participants will wear three accelerometers on their wrists and right hip to monitor the minutes of exercise, postural change, activity counts and energy expenditure for exploration during the whole 2-hour session, one session/each week for 12 weeks. An activity log will be applied to record the driving and play duration, driving locations, and the caregiver's feedback on the training program every week. All videotapes will be coded by two independent coders.

Intervention: The research team will ask caregivers to identify goals (before intervention), and measure progress using goal-attainment scaling (GAS) at T1 and T2 time points for the four groups. The training principles are similar to those applied in our previous studies of ROC training in various environments. To record the total driving time, locations, and caregivers' feedback regarding training, an activity log will be used for each session. All groups will continue their regular therapy throughout the 24-week duration of the study, including physical therapy, occupational therapy, and speech therapy.

Follow-up: This period will involve 12-weeks following the above treatment programs; during this time no treatment programs will be delivered to the participants except for their own regular therapy.

Instrument and Procedure: To present a complete investigation of participants' changes on the 3 domains of ICF, home affordances and parenting stress levels, the investigators will provide standardized assessments as the quantitative measures at T1, T2, and T3, and behavioral observations and activity logs as the qualitative measures during the intervention. In addition, accelerometers will be applied during the intervention to provide a quantitative measure for exploration, including the minutes of exercise, postural change, activity counts and energy expenditure.

Data Reduction and Analysis Quantitative measures at T1, T2, and T3 Repeated measure one way ANOVA will be used to compare the mean difference of using different toy cars on mobility, socialization and exploratory behaviors before and after the intervention, and after 12-week follow-up, i.e., within group comparison. One way ANOVA will be used to compare the mean difference of all developmental tests, participation and physical activity for exploration among three groups before and after the intervention and the end of follow-up phase.

Descriptive statistics including frequency, means, standard deviations, as well as nonparametric data medians and interquartile ranges will be calculated. Data will be analyzed based on an intention-to-treat analysis. A repeated measures analysis of variance (group [4] × time [3]) will be employed to evaluate the treatment effects on the primary and secondary outcomes among the 4 groups at T1, T2, and T3, followed by a post-hoc analysis using Bonferroni test to determine between which groups the differences occur.

Descriptive statistics (frequency, means, standard deviations) of each behavior will be calculated and repeated measures analysis of variance (group [4] × time [12]) will be used to compare the effects of behavioral measures among the 4 groups during intervention. Furthermore, the quantitative data obtained from the accelerometers during intervention will be organized and calculated. A repeated measures analysis of variance (group [4] × time [12]) will also be used to compare the effects related to exploration among the 4 groups during intervention.

ELIGIBILITY:
Inclusion Criteria:

1. motor delays that resulted in motor impairments that prevented independent walking (standard deviation (SD) > 1.5, assessed by the Chinese Child Development Inventory59,60 via a pediatric physician)
2. can stand independently for two seconds or to tolerate standing with support for 10 minutes
3. can reach objects with either one or two hands
4. the height is between 69 to 103 cm and the weight is between 7-18 kg
5. parents are able to provide consent for their child's participation in the ROC training programs.

Exclusion Criteria:

1. children with severe sensory impairments such as blindness, deafness
2. the height is not between 69 to 103 cm and the weight is not between 7 to 18 kg
3. parents/caregivers are not able to make a time commitment for the training phase

Ages: 1 Year to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 19 (Actual)
Dates: Start 2018-11-15 (Actual); Primary Completion 2020-06-28 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Mobility and Social Function at 12 Weeks | PEDI will be administered on two occasions: before and after the 12-week intervention (T1 & T2).
  The Chinese version of Pediatric Evaluation of Disability Inventory (PEDI-C) is a set of tests for children from 8 months to 6 years old. The PEDI-C quantifies self-care, mobility, and social function, and is particularly useful for tracking changes in functional skills. Each domain can be used separately for data analysis. The inter-rater and intra-rater reliabilities of the study reveal excellent agreement of the observations (0.95-0.99), and good concurrent validity with the Functional Independence Measure for Children (Spearman ρ, 0.92-0.99).
Mobility-Driving Performance | 30 minutes/per week for a total of 12 weeks
  Every week during the intervention phase, the 70-minute driving will be recorded and the most active 30 minutes will be selected for coding. The following behaviors will be coded, including driving categories (independent mobility, assisted mobility, caregiver mobility), visual attention to the switch and stopping categories (independent stop, stops with verbal cues, stops with tactile contacts).
Socialization | 40 minutes/per week for a total of 12 weeks
  The behaviors of social interactions are obtained during the most active 30 minutes of driving and the most active 10 minutes of the recorded 20-minute natural play, i.e., the first 20 minutes of natural play. From these videotapes, the frequency and duration of the following will be coded: physical contacts, initiation of contact with others, other initiated contacts, facial expressions, vocalizations/gestures and mutual play events (e.g. sharing an object or a toy).
Change from Posttest Mobility and Social Function at 12 Weeks | PEDI will be administered on two occasions: after the 12-week intervention (T2) and the end of the 12-week follow-up phase (T3).
  The Chinese version of Pediatric Evaluation of Disability Inventory (PEDI-C) is a set of tests for children from 8 months to 6 years old. The PEDI-C quantifies self-care, mobility, and social function, and is particularly useful for tracking changes in functional skills. Each domain can be used separately for data analysis. The inter-rater and intra-rater reliabilities of the study reveal excellent agreement of the observations (0.95-0.99), and good concurrent validity with the Functional Independence Measure for Children (Spearman ρ, 0.92-0.99).

SECONDARY OUTCOMES:
Change from Baseline Sit-to-Stand at 12 Weeks | This test will be administered on two occasions: before and after the 12-week intervention (T1 & T2).
  5-repetition Sit-to-stand (STS) is a body function test measures the time required to complete five consecutive sit-to-stand cycles as quickly as possible as timed by a stopwatch. Participants will be tested barefoot on a firm mat and the starting position with hip flexed at 90 degrees and knee flexed at 105 degrees. The intraclass correlation coefficients of intra-session reliability and test-retest reliability were 0.95 and 0.99 respectively. The convergent validity was supported by significant correlation with isometric muscle strength, scores of Gross Motor Function Measure, and gait function (r or rho = 0.45-0.78).
Change from Posttest Sit-to-Stand at 12 Weeks | This test will be administered on two occasions: after the 12-week intervention (T2) and the end of the 12-week follow-up phase (T3).
  5-repetition Sit-to-stand (STS) is a body function test measures the time required to complete five consecutive sit-to-stand cycles as quickly as possible as timed by a stopwatch. Participants will be tested barefoot on a firm mat and the starting position with hip flexed at 90 degrees and knee flexed at 105 degrees. The intraclass correlation coefficients of intra-session reliability and test-retest reliability were 0.95 and 0.99 respectively. The convergent validity was supported by significant correlation with isometric muscle strength, scores of Gross Motor Function Measure, and gait function (r or rho = 0.45-0.78).
Change from Baseline Mastery Motivation at 12 Weeks | This test will be administered on two occasions: before and after the 12-week intervention (T1 & T2).
  The Revised Dimensions of Mastery Questionnaire (DMQ 18)-Chinese version is a body function test and used to measure mastery motivation through caregivers' report. The DMQ has 7 scales: cognitive/object persistence, gross motor persistence, social mastery motivation with adults, social mastery motivation with children/peers, mastery pleasure, negative reactions to challenge in mastery situations, and general competence. A Likert-type scale of 1-5 is used to rate the similarity; lower score indicates lower similarity. The DMQ 18 has four parallel age-related versions for children aged 6 months to 19 years (infant, preschool, school-age rated by adults, and school-age self-report). We utilized the infant version (approximately 6-23 months) and preschool version (approximately 2-6 years) according to the age of the participants. The DMQ 18 shows good validity, internal consistency, and acceptable intra- and inter-rater reliability.
Change from Posttest Mastery Motivation at 12 Weeks | This test will be administered on two occasions: after the 12-week intervention (T2) and the end of the 12-week follow-up phase (T3).
  The Revised Dimensions of Mastery Questionnaire (DMQ 18)-Chinese version is a body function test and used to measure mastery motivation through caregivers' report. The DMQ has 7 scales: cognitive/object persistence, gross motor persistence, social mastery motivation with adults, social mastery motivation with children/peers, mastery pleasure, negative reactions to challenge in mastery situations, and general competence. A Likert-type scale of 1-5 is used to rate the similarity; lower score indicates lower similarity. The DMQ 18 has four parallel age-related versions for children aged 6 months to 19 years (infant, preschool, school-age rated by adults, and school-age self-report). We utilized the infant version (approximately 6-23 months) and preschool version (approximately 2-6 years) according to the age of the participants. The DMQ 18 shows good validity, internal consistency, and acceptable intra- and inter-rater reliability.
Change from Baseline Developmental Abilities at 12 Weeks | This test will be administered on two occasions: before and after the 12-week intervention (T1 & T2).
  The Bayley Scales of Development (Bayley) is an internationally recognized set of developmental tests that involve play and parental questionnaires. The Bayley has subsets of tests for motor (fine and gross), language (receptive and expressive), and cognitive development, ages from 0-3 years old. The intra- and inter-rater reliability were high for the Bayley III (ICCs=0.88-0.99 and SEMs=0.59-1.60). For discriminative validity, term infants scored significantly higher than preterm infants on the Bayley II and III cognitive (effect size=0.36-0.92 vs. 0.55-0.62), language (effect size=0.20-0.50 vs. 0.22-0.37), and motor scales (effect size=0.48-0.70 vs. 0.48-0.67) over age (all p<0.05).
Change from Posttest Developmental Abilities at 12 Weeks | This test will be administered on two occasions: after the 12-week intervention (T2) and the end of the 12-week follow-up phase (T3).
  The Bayley Scales of Development (Bayley) is an internationally recognized set of developmental tests that involve play and parental questionnaires. The Bayley has subsets of tests for motor (fine and gross), language (receptive and expressive), and cognitive development, ages from 0-3 years old. The intra- and inter-rater reliability were high for the Bayley III (ICCs=0.88-0.99 and SEMs=0.59-1.60). For discriminative validity, term infants scored significantly higher than preterm infants on the Bayley II and III cognitive (effect size=0.36-0.92 vs. 0.55-0.62), language (effect size=0.20-0.50 vs. 0.22-0.37), and motor scales (effect size=0.48-0.70 vs. 0.48-0.67) over age (all p<0.05).
Change from Baseline Home Affordances at 12 Weeks | This test will be administered on two occasions: before and after the 12-week intervention (T1 & T2).
  The Affordances in the Home Environment for Motor Development (AHEMD) is a reliable and valid assessment to assess the quality and quantity of motor development opportunities in the home during early childhood. Age-related AHEMD questionnaires were developed (3-to-18 months; and 18-to-42 months) and translated into four different languages: English, Chinese, Portuguese, and Spanish. Test-retest reliabilities for AHEMD-Toddler-C were adequate (0.46~0.93). For convergent validity, the correlation coefficients between AHEMD and HOME were 0.44.
Change from Posttest Home Affordances at 12 Weeks | This test will be administered on two occasions: after the 12-week intervention (T2) and the end of the 12-week follow-up phase (T3).
  The Affordances in the Home Environment for Motor Development (AHEMD) is a reliable and valid assessment to assess the quality and quantity of motor development opportunities in the home during early childhood. Age-related AHEMD questionnaires were developed (3-to-18 months; and 18-to-42 months) and translated into four different languages: English, Chinese, Portuguese, and Spanish. Test-retest reliabilities for AHEMD-Toddler-C were adequate (0.46~0.93). For convergent validity, the correlation coefficients between AHEMD and HOME were 0.44.
Change from Baseline Goal Achievements at 12 Weeks | This test will be administered on two occasions: before and after the 12-week intervention (T1 & T2).
  Goal Attainment Scale (GAS) is a family-centered, criterion-referenced and responsive tool. There are 5 possible outcomes: a score of 0 means the child has attained the goal, whereas scores of -2 and -1 represent lower than expected performance and +1 and +2 are higher than expected performance. Level of satisfaction with goal achievement was also assessed by parents on a weekly basis using a 5-point. Likert scale: 1=very satisfied, 2=somewhat satisfied, 3=neither satisfied nor unsatisfied, 4=somewhat unsatisfied, 5=very unsatisfied. It has excellent inter-rater agreements with inter-class correlations of 0.90 or above. GAS was shown to correlate strongly with other measures that showed change, and it discriminated between lower and higher functional or QOL status.
Change from Posttest Goal Achievements at 12 Weeks | This test will be administered on two occasions: after the 12-week intervention (T2) and the end of the 12-week follow-up phase (T3).
  Goal Attainment Scale (GAS) is a family-centered, criterion-referenced and responsive tool. There are 5 possible outcomes: a score of 0 means the child has attained the goal, whereas scores of -2 and -1 represent lower than expected performance and +1 and +2 are higher than expected performance. Level of satisfaction with goal achievement was also assessed by parents on a weekly basis using a 5-point. Likert scale: 1=very satisfied, 2=somewhat satisfied, 3=neither satisfied nor unsatisfied, 4=somewhat unsatisfied, 5=very unsatisfied. It has excellent inter-rater agreements with inter-class correlations of 0.90 or above. GAS was shown to correlate strongly with other measures that showed change, and it discriminated between lower and higher functional or QOL status.
Change from Baseline Parental Stress at 12 Weeks | This test will be administered on two occasions: before and after the 12-week intervention (T1 & T2).
  Parental Perceptions-Parenting Stress Index (PSI) is a tool that was designed to measure the overall level of parenting stress experienced by parents of children between the ages of 1 month and 12 years. PSI was also translated into Chinese language (PSI-C) and showed very god reliability (from parent : .55-.80). The validity was well established (factorial validity: 41% of variance on child section accounted for by 6 factors; 44% on Parent section by 7 parent factors).
Change from Posttest Parental Perceptions at 12 Weeks | This test will be administered on two occasions: after the 12-week intervention (T2) and the end of the 12-week follow-up phase (T3).
  Parental Perceptions is a set of self-developed questionnaires from the previous studies, which will also be used at T1, T2 and T3 to provide examine parental perceptions on the PMDs use and children's capabilities.
Energy expenditure for Exploration | 2 hours each week for a total of 12 weeks
  Each week the participant wears the accelerometers (ActiGraph®GT9X) on each wrist and right hip during the 2-hour training session, one session/ peer week. The accelerometers code the energy expenditure and physical activity for driving and playing. Combining with the results from the activity logs and videotapes, this data enables us to monitor the energy expenditure, minutes of exercise, postural change, and activity counts for exploration.

CONTACTS AND LOCATIONS:
Overall Officials: Hsiang-Han Huang, ScD, Principal Investigator — Chang Gung University
Locations (2):
- Taiwan (2):
  - Chang Gung University, Taoyuan, Taoyuan County
  - Linkou Chang Gung Memorial Hospital, Taoyuan, Taoyuan County

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Huang HH, Chu YW, Chan AT, Chen CL. A pilot randomised controlled trial of ride-on cars and postural combinations of standing and sitting for mobility and social function in toddlers with motor delays. Disabil Rehabil Assist Technol. 2025 Jan;20(1):53-63. doi: 10.1080/17483107.2023.2299712. Epub 2024 Jan 5. PMID 38180348